CLINICAL TRIAL: NCT00224406
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Repertaxin in the Prevention of Primary Graft Dysfunction After Lung Transplantation
Brief Title: Repertaxin in Prevention of Primary Graft Dysfunction After Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REP0104
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Ischemia-Reperfusion Injury; Lung Transplantation
Keywords: Lung transplantation; Reperfusion Injury; Survival
MeSH Terms: conditions — Reperfusion Injury | interventions — reparixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All personnel involved and patients participating in the study were to remain blinded to the patient randomization codes with the exception of those involved in packaging and labelling the study medication. After the database lock of data recorded in the main part of the study, corresponding to the Month 1 follow-up visit of the last patient in, the blind code was broken and the study continued in an open fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Repertaxin (Experimental): Both repertaxin and placebo were aqueous solutions packaged into identical clear glass Type I ampoule single dose units. Each ampoule contained 10 mL of either repertaxin or placebo.The dosing solution for infusion was prepared aseptically at the designated Pharmacy within each center and dispensed as 12.65 mg/mL solution in appropriate size infusion bags. An initial 'loading dose' of Repertaxin of 4.488 mg/kg body weight/hour was administered over 30 minutes followed by a maintenance dose of 2.772 mg/kg body weight/hour lasting 47.5 hours.The loading and maintenance doses were administered using the same dosing solution (Repertaxin 12.65 mg/ml), but with the pump rate altered to provide an infusion rate of approximately 0.35 mUkg/hour and 0.22 ml/kg/hour, respectively.
  Interventions: Drug: Repertaxin
- Placebo (Placebo Comparator): Both repertaxin and placebo were aqueous solutions packaged into identical clear glass Type I ampoule single dose units. The dosing solution for infusion was prepared aseptically at the designated Pharmacy within each center and dispensed as 12.65 mg/mL solution in appropriate size infusion bags. ampoule contained 10 mL of either repertaxin or placebo. An initial 'loading dose' of 9 mg/ml sodium chloride (NaCl) solution was administered over 30 minutes, followed by a maintenance dose lasting 47.5 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Repertaxin — An initial 'loading dose' of repertaxin was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The study medication was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
  Arms: Repertaxin
Other: Placebo — An initial 'loading dose' of placebo was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The placebo was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
The objective of this clinical study was to evaluate whether CXCL8 (CXC ligand 8 [formerly interleukin (IL)-8]) inhibition with repertaxin leads to reduced severity of primary graft dysfunction, as the result of improved functional and clinical outcomes in lung transplantation patients.

The safety of repertaxin in the specific clinical setting was also evaluated.

The ability of repertaxin to reduce target cells (polymorphonuclear leukocyte [PMN]) infiltration into the graft was evaluated to confirm its mechanism of action.

DETAILED DESCRIPTION:
This was a phase 2, multi-center, randomized, double-blind, placebo-controlled, parallel-group (two arms) study.

A total of 100 patients accepted and listed for lung transplantation, who met all of the study inclusion and none of the exclusion criteria described in Sections 9.3.1 and 9.3.2 of this report, were planned to be enrolled in the study. These patients were randomly assigned in a 1:1 ratio to receive either repertaxin or placebo, by continuous intravenous infusion for a period of 48 hours to start approximately 2 hours before reperfusion of the (first) transplanted lung occurred.

The experimental treatment was additional to the standard treatment of lung transplant recipients.

An initial 'loading dose' of repertaxin of 4.488 mg/kg body weight/hour was to be administered over 30 minutes followed by a maintenance dose of 2.772 mg/kg body weight/hour lasting 47.5 hours.

Placebo was to be volume matched saline. Total infusion volume was not to exceed 500 mL/24 hours. Study medication was to be provided as clear glass class I ampoules, each containing 10 mL of the following products: repertaxin (33 mg/mL aqueous injectable solution) and placebo (9 mg/mL aqueous injectable solution of NaCl).

The double-blind was to be maintained for the main part of the study only, i.e. up to the Month 1 (at least 30 days post-transplant) follow-up visit of the last patient in. After database lock of Month 1 data the study proceeded in an open fashion.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted and listed for transplantation due to irreversible, progressive disabling, end-stage pulmonary disease;
* Ages 18 to 65 years;
* Body weight 30 to 95 kg (inclusive) (i.e. up to 95.99 kg);
* Planned isolated (single and bi-lateral) lung transplant from a non-living donor with brain death. This included lobar lung transplant involving excision and sizing of a cadaver donor lobe to meet the thoracic dimension of the recipient before being transplanted;
* Normal renal function at the time of transplant as per calculated creatinine clearance (Clcr) 60 mL/min. Creatinine clearance was calculated according to the Cockcroft-Gault formula;
* Patient was willing and able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations;
* Patient gave written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent could be withdrawn by the patient at any time without prejudice to their future medical care.

Exclusion Criteria:

* Recipients of an intended multiple organ transplant, including heart-lung and liver-lung transplantation;
* Recipients of a lung from a living lobar donor;
* Recipients of a lung from a non-heart beating donor;
* Re-do lung transplantation;
* Recipients requiring mechanical ventilation at the time of transplant;
* Recipients with an extra-respiratory tract site of infection (positive blood culture(s) and/or fever associated with other signs of systemic sepsis syndrome). The criterion was not meant to exclude bacteraemic cystic fibrosis patients with or without fever, unless they presented with other signs of sepsis;
* Recipients with hepatic dysfunction (bilirubin exceeding 3 mg/dL and/or transaminases >3X upper limit of normal [ULN]) at the time of transplant;
* Hypersensitivity to:

  * Ibuprofen or to more than one non steroidal anti-inflammatory drug (NSAID);
  * Medications belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib;
* Patients simultaneously participating in any other studies involving a study drug to be administered concomitantly with the investigational product and/or a study drug intended to prevent ischemia/reperfusion injury;
* Planned use of anli-CD3 monoclonal antibody (Orthoclone OKT3) or alemtuzumab (Campath) induction immunosuppression;
* Planned use of sirolimus in the first 3 months after transplantation;
* Pregnant or breast-feeding women (NB: pregnancy was lo be avoided in patients or partners during the first month of participation in the study; no other specific warnings were described, considering even stricter general recommendations concerning pregnancy in transplanted patients, the treatment course of the investigational product, its pharmacokinetic profile, and the lack of significant adverse effects on mating performance and fertility in animal studies).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2006-09-13 (Actual); Study Completion 2007-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Novellini, MD, Study Director — Dompé Farmaceutici S.p.A
Locations (6):
- United States (5):
  - University of South California, Department of Cardiothoracic Surgery, Los Angeles, California
  - University of Colorado, Health Sciences Centre, Denver, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
- Toronto General Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 233 subjects were screened, of whom 114 were randomised and 119 were screen failures.
Pre-assignment Details: In total 114 subjects were randomised 1:1 to Repertaxin or Placebo, with slightly more assigned to the Placebo group (59 compared to 55 Repertaxin). 101 patients received study drug and were included in the ITT and safety population (46 on Repertaxin; 55 on placebo).
Groups:
- Repertaxin: An initial 'loading dose' of Repertaxin of 4.488 mg/kg body weight/hour was administered over 30 minutes followed by a maintenance dose of 2.772 mg/kg body weight/hour lasting 47.5 hours.The loading and maintenance doses were administered using the same dosing solution (Repertaxin 12.65 mg/ml), but with the pump rate altered to provide an infusion rate of approximately 0.35 mUkg/hour and 0.22 ml/kg/hour, respectively.
  Repertaxin: An initial 'loading dose' of repertaxin was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The study medication was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
- Placebo: An initial 'loading dose' of 9 mg/ml sodium chloride (NaCl) solution was administered over 30 minutes, followed by a maintenance dose lasting 47.5 hours.
  Placebo: An initial 'loading dose' of placebo was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The placebo was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
Period: Overall Study
Arm/Group | Repertaxin | Placebo
Started | 55 | 59
Intention to Treat Population (ITT) | 46 | 55
Per Protocol Population (PP) | 46 | 53
Safety Population (SAF) | 46 | 55
Completed | 46 | 52
Not Completed | 9 | 7
Not completed — Re-transplant | 0 | 2
Not completed — Death | 0 | 1
Not completed — Transplant cancelled | 0 | 4
Not completed — Drug not delivered | 2 | 0
Not completed — Other | 4 | 0
Not completed — Transplant cancelled | 3 | 0

BASELINE CHARACTERISTICS:
Population: The safety population (SAF) consisted of all patients who received any study medication and was based on the treatment actually received.
Groups:
- Repertaxin (SAF): Both repertaxin and placebo were aqueous solutions packaged into identical clear glass Type I ampoule single dose units. Each ampoule contained 10 mL of either repertaxin or placebo.The dosing solution for infusion was prepared aseptically at the designated Pharmacy within each center and dispensed as 12.65 mg/mL solution in appropriate size infusion bags. An initial 'loading dose' of Repertaxin of 4.488 mg/kg body weight/hour was administered over 30 minutes followed by a maintenance dose of 2.772 mg/kg body weight/hour lasting 47.5 hours.The loading and maintenance doses were administered using the same dosing solution (Repertaxin 12.65 mg/ml), but with the pump rate altered to provide an infusion rate of approximately 0.35 mUkg/hour and 0.22 ml/kg/hour, respectively.
  Repertaxin: An initial 'loading dose' of repertaxin was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The study medication was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
- Placebo (SAF): Both repertaxin and placebo were aqueous solutions packaged into identical clear glass Type I ampoule single dose units. The dosing solution for infusion was prepared aseptically at the designated Pharmacy within each center and dispensed as 12.65 mg/mL solution in appropriate size infusion bags. ampoule contained 10 mL of either repertaxin or placebo. An initial 'loading dose' of 9 mg/ml sodium chloride (NaCl) solution was administered over 30 minutes, followed by a maintenance dose lasting 47.5 hours.
  Placebo: An initial 'loading dose' of placebo was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The placebo was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
- Total: Total of all reporting groups
Arm/Group | Repertaxin (SAF) | Placebo (SAF) | Total
Number analyzed (Participants) | 46 | 55 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 46 | 50 | 96
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.5) | 50.9 (12.2) | 48.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 23 | 28 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 45 | 55 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 17 | 33
  United States | 30 | 38 | 68

OUTCOME MEASURES:

1. Primary Outcome: PaO2/FiO2 Ratio at ICU Admission (Time 0) and 24 Hours
Description: The PaO2/FiO2 ratio was calculated to assess the severity of hypoxemia, or low blood oxygen levels. A low PaO2/FiO2 value has been associated with increased mortality and hospital stay in patients admitted to the intensive care unit (ICU). It was calculated by dividing the partial pressure of oxygen in arterial blood (PaO2) by the fraction of inspired oxygen (FiO2). A normal P/F ratio was typically above 300, and a lower ratio indicates a greater severity of hypoxemia. As the Pa02/Fi02 ratio was dependent on altitude, data were corrected for altitude in the analyses of corrected data. The correction factor is defined as (Pressure at Denver)/(Pressure at sea level) = 633/760 = 0.8329; PaO2 values were corrected as follows: Corrected value = measured value/0.8329
Time Frame: At T0 (time of ICU admission) and 24 hours post-ICU admission
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Mean (Standard Deviation); unit: ratio of PaO2/FiO2
Groups:
- Repertaxin (ITT): Both repertaxin and placebo were aqueous solutions packaged into identical clear glass Type I ampoule single dose units. Each ampoule contained 10 mL of either repertaxin or placebo.The dosing solution for infusion was prepared aseptically at the designated Pharmacy within each center and dispensed as 12.65 mg/mL solution in appropriate size infusion bags. An initial 'loading dose' of Repertaxin of 4.488 mg/kg body weight/hour was administered over 30 minutes followed by a maintenance dose of 2.772 mg/kg body weight/hour lasting 47.5 hours.The loading and maintenance doses were administered using the same dosing solution (Repertaxin 12.65 mg/ml), but with the pump rate altered to provide an infusion rate of approximately 0.35 mUkg/hour and 0.22 ml/kg/hour, respectively.
  Repertaxin: An initial 'loading dose' of repertaxin was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The study medication was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
- Placebo (ITT): Both repertaxin and placebo were aqueous solutions packaged into identical clear glass Type I ampoule single dose units. The dosing solution for infusion was prepared aseptically at the designated Pharmacy within each center and dispensed as 12.65 mg/mL solution in appropriate size infusion bags. ampoule contained 10 mL of either repertaxin or placebo. An initial 'loading dose' of 9 mg/ml sodium chloride (NaCl) solution was administered over 30 minutes, followed by a maintenance dose lasting 47.5 hours.
  Placebo: An initial 'loading dose' of placebo was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The placebo was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
ratio of PaO2/FiO2
  ICU Admission (Time 0) | 346.3 (125.5) | 337.9 (143.0)
  24 Hours Post ICU Admission: number analyzed (Participants) | 24 | 29
  24 Hours Post ICU Admission | 320.1 (119.5) | 307.3 (111.3)
Statistical Analysis 1: Comparison: Repertaxin (ITT) vs Placebo (ITT); Repeated Measurements Analysis of PaO2/FiO2 ratio corrected for the altitude at 0 and 24hours after ICU admission using a one-sided test excluding missing data. Herein analysis at ICU Admission (Time 0); Test type: Superiority; p = 0.8541, t-test, 1 sided; Mean Difference (Final Values) = 5.022, 95% CI 1-sided [upper limit 50.26]
Statistical Analysis 2: Comparison: Repertaxin (ITT) vs Placebo (ITT); Repeated Measurements Analysis of PaO2/FiO2 ratio corrected for the altitude at 0 and 24hours after ICU admission using a one-sided test excluding missing data. Herein analysis at 24 Hours Post ICU Admission; Test type: Superiority; p = 0.6996, t-test, 1 sided; Mean Difference (Final Values) = 10.426, 95% CI 1-sided [upper limit 55.17]

2. Secondary Outcome: PaO2/FiO2 Ratio (ICU Admission Then 24 Hours up to Extubation or up to 72 Hours)
Description: Time profile of oxygenation was a comparison of the sequential measurements of the ratios of arterial PaO2 to inspired oxygen fractions FiO2. Herein repeated measurements analysis of PaO2/FiO2 ratio corrected after ICU admission using a one-sided test excluding missing data.
Time Frame: At ICU admission (T0), 24, 48 and 72 hours post-ICU admission
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Mean (Standard Deviation); unit: ratio of PaO2/FiO2
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
ratio of PaO2/FiO2
  ICU Admission (Time 0) | 346.3 (125.5) | 337.9 (143.0)
  24 Hours Post ICU Admission: number analyzed (Participants) | 24 | 29
  24 Hours Post ICU Admission | 320.1 (119.5) | 307.3 (111.3)
  48 Hours Post ICU Admission: number analyzed (Participants) | 14 | 17
  48 Hours Post ICU Admission | 266.1 (117.3) | 279.2 (151.8)
  72 Hours Post ICU Admission: number analyzed (Participants) | 12 | 10
  72 Hours Post ICU Admission | 275.6 (88.1) | 233.9 (132.0)
Statistical Analysis 1: Comparison: Repertaxin (ITT) vs Placebo (ITT); ICU Admission (Time 0); Test type: Superiority; p = 0.8654, t-test, 1 sided; Mean Difference (Final Values) = 4.377, 95% CI 1-sided [upper limit 47.15]
Statistical Analysis 2: Comparison: Repertaxin (ITT) vs Placebo (ITT); 24 Hours Post ICU Admission; Test type: Superiority; p = 0.6789, t-test, 1 sided; Median Difference (Final Values) = 13.386, 95% CI 1-sided [upper limit 66.91]
Statistical Analysis 3: Comparison: Repertaxin (ITT) vs Placebo (ITT); 48 Hours Post ICU Admission; Test type: Superiority; p = 0.6345, t-test, 1 sided; Mean Difference (Final Values) = -19.968, 95% CI 1-sided [upper limit 49.56]
Statistical Analysis 4: Comparison: Repertaxin (ITT) vs Placebo (ITT); 72 Hours Post ICU Admission; Test type: Superiority; p = 0.9858, t-test, 1 sided; Mean Difference (Final Values) = 0.908, 95% CI 1-sided [upper limit 85.49]

3. Secondary Outcome: Number of Patients With Different Primary Graft Dysfunction (PGD) Scores (0-3, and Missing Data)
Description: PGD after lung transplantation ranged from mild to severe depending on the level of hypoxaemia and lung injury post-transplant.
  PGD score was calculated according to the scoring system below:
  Grade 0 PaO2/FiO2 >=300 mmHg; no radiographic infiltrates (RI); Grade 1 PaO2/FiO2 >=300mmHg + RI consistent with pulmonary oedema; Grade 2 200 mmHg <=PaO2/FiO2 <=300 mm Hg + RI consistent with pulmonary oedema; Grade 3 PaO2/FiO2 < 200 mm Hg + RI consistent with pulmonary oedema. The higher the score, the worse the outcome. Any patient with no infiltrate on chest X-rays was automatically Grade 0. If the patient was on nasal cannula for oxygen or FiO2 <0.3, the patient was graded as 0 or 1, based on chest X-rays. Any patient on extracorporeal membrane oxygenation was Grade 3. Any subject mechanically ventilated with FiO2 greater than 0.5 or requiring nitric oxide beyond 48 hours from the time of transplant was Grade 3.
Time Frame: At ICU admission (T0), 24, 48 and 72 hours post-ICU admission
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
Participants
  ICU Admission (Time 0) - PGD Score Missing | 0 | 1
  ICU Admission (Time 0) - PGD Score 0 | 28 | 33
  ICU Admission (Time 0) - PGD Score 1 | 9 | 8
  ICU Admission (Time 0) - PGD Score 2 | 6 | 4
  ICU Admission (Time 0) - PGD Score 3 | 3 | 9
  24 Hours Post ICU Admission - PGD Score Missing | 0 | 1
  24 Hours Post ICU Admission - PGD Score 0 | 22 | 30
  24 Hours Post ICU Admission - PGD Score 1 | 14 | 12
  24 Hours Post ICU Admission - PGD Score 2 | 5 | 6
  24 Hours Post ICU Admission - PGD Score 3 | 5 | 6
  48 Hours Post ICU Admission - PGD Score Missing | 0 | 3
  48 Hours Post ICU Admission - PGD Score 0 | 22 | 24
  48 Hours Post ICU Admission - PGD Score 1 | 15 | 17
  48 Hours Post ICU Admission - PGD Score 2 | 4 | 2
  48 Hours Post ICU Admission - PGD Score 3 | 5 | 9
  72 Hours Post ICU Admission - PGD Score Missing | 1 | 3
  72 Hours Post ICU Admission - PGD Score 0 | 22 | 27
  72 Hours Post ICU Admission - PGD Score 1 | 16 | 17
  72 Hours Post ICU Admission - PGD Score 2 | 3 | 2
  72 Hours Post ICU Admission - PGD Score 3 | 4 | 6
Statistical Analysis 1: Comparison: Repertaxin (ITT) vs Placebo (ITT); Analysis of PGD score was performed separately at time 0, and at 24, 48, 72 hours after ICU admission. Herein analysis at ICU Admission (Time 0). One patient of placebo group is excluded from analysis of PGD score because the cause of graft dysfunction is Cardiogenic pulmonary edema; Test type: Superiority; p = 0.7985, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.867, 95% CI 2-sided [0.727 to 11.302] — Odds ratio is Repertaxin:Placebo ratio of PGD scores 0-2:PGD score 3 odds
Statistical Analysis 2: Comparison: Repertaxin (ITT) vs Placebo (ITT); Analysis of PGD score was performed separately at time 0, and at 24, 48, 72 hours after ICU admission. Herein analysis at 24h post-ICU admission. One patient of placebo group is excluded from analysis of PGD score because the cause of graft dysfunction is Cardiogenic pulmonary edema; Test type: Superiority; p = 0.5606, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.837, 95% CI 2-sided [0.226 to 3.092] — Odds ratio is Repertaxin:Placebo ratio of PGD scores 0-2:PGD score 3 odds
Statistical Analysis 3: Comparison: Repertaxin (ITT) vs Placebo (ITT); Analysis of PGD score was performed separately at time 0, and at 24, 48, 72 hours after ICU admission. Herein analysis at 48h post-ICU admission. One patient of placebo group is excluded from analysis of PGD score because the cause of graft dysfunction is Cardiogenic pulmonary edema; Test type: Superiority; p = 0.8786, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.716, 95% CI 2-sided [0.531 to 5.552] — Odds ratio is Repertaxin:Placebo ratio of PGD scores 0-2:PGD score 3 odds
Statistical Analysis 4: Comparison: Repertaxin (ITT) vs Placebo (ITT); Analysis of PGD score was performed separately at time 0, and at 24, 48, 72 hours after ICU admission. Herein analysis at 72h post-ICU admission. One patient of placebo group is excluded from analysis of PGD score because the cause of graft dysfunction is Cardiogenic pulmonary edema; Test type: Superiority; p = 0.8499, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.337, 95% CI 2-sided [0.352 to 5.072] — Odds ratio is Repertaxin:Placebo ratio of PGD scores 0-2:PGD score 3 odds

4. Secondary Outcome: Time to Freedom From Mechanical Ventilation
Description: Time to freedom from mechanical ventilation was defined as "time between admission to the ICU and the initial time of first extubation (breathing off mechanical ventilation without a tube) which was maintained for more than 24 hours". This number was measured in hours and was derived as (date/time of extubation-date/time of ICU admission)/3600. The longer the time, the worst the outcome.Time to freedom from mechanical ventilation, if greater than 1 month (720 hours), was censored to 720 hours. Patients re-transplanted were censored at the date/time of re-transplant. Herein differences in the time to freedom from mechanical ventilation were reported between placebo and repertaxin.
Time Frame: At 24, 48, 72 hours post ICU admission
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
hours
  24 Hours Post-ICU Admission: number analyzed (Participants) | 23 | 28
  24 Hours Post-ICU Admission | 0.5000 (0.0737) | 0.4909 (0.0674)
  48 Hours Post-ICU Admission: number analyzed (Participants) | 14 | 15
  48 Hours Post-ICU Admission | 0.6957 (0.0678) | 0.7273 (0.0601)
  72 Hours Post-ICU Admission: number analyzed (Participants) | 12 | 10
  72 Hours Post-ICU Admission | 0.7391 (0.0647) | 0.8052 (0.0541)
Statistical Analysis 1: Comparison: Repertaxin (ITT) vs Placebo (ITT); Test type: Superiority — at 24 hrs from mechanical ventilation; p = 0.7076, Log Rank; difference in event probability = 0.0091, 95% CI 2-sided [-0.1867 to 0.2049]
Statistical Analysis 2: Comparison: Repertaxin (ITT) vs Placebo (ITT); at 48 hrs from mechanical ventilation; Test type: Superiority; p = 0.7076, Log Rank; difference in event probability = -0.0316, 95% CI 2-sided [-0.2092 to 0.1460]
Statistical Analysis 3: Comparison: Repertaxin (ITT) vs Placebo (ITT); at 72 hrs from mechanical ventilation; Test type: Superiority; p = 0.7076, Log Rank; difference in event probability = -0.0661, 95% CI 2-sided [-0.2314 to 0.0993]

5. Secondary Outcome: Probability of Death During Intensive Care Unit (ICU) Stay at Different Timepoints
Description: The duration of ICU stay, in term of hours, at different timepoints, in both placebo and repertaxin groups, was measured. The longer the ICU stay, the worse the outcome. mean event probability" (death) and its standard error (SE) at each timepoint.
Time Frame: At 24, 48, 72 hours post ICU admission
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Mean (Standard Error); unit: event probability
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
event probability
  At 24 h hours post ICU admission: number analyzed (Participants) | 46 | 53
  At 24 h hours post ICU admission | 0.0000 (0.0000) | 0.0364 (0.0252)
  At 48 h hours post ICU admission: number analyzed (Participants) | 31 | 39
  At 48 h hours post ICU admission | 0.3261 (0.0691) | 0.2909 (0.0612)
  At 72 h hours post ICU admission: number analyzed (Participants) | 24 | 27
  At 72 h hours post ICU admission | 0.4783 (0.0737) | 0.4962 (0.0679)
Statistical Analysis 1: Comparison: Repertaxin (ITT) vs Placebo (ITT); Analysis at 24 hours; Test type: Superiority; p = 0.9632, Log Rank; Difference in event probability = -0.0364, 95% CI 2-sided [-0.0858 to 0.0131]
Statistical Analysis 2: Comparison: Repertaxin (ITT) vs Placebo (ITT); Analysis at 48 h; Test type: Superiority; p = 0.9632, Log Rank; Difference in event probability = 0.0352, 95% CI 2-sided [-0.1458 to 0.2162]
Statistical Analysis 3: Comparison: Repertaxin (ITT) vs Placebo (ITT); analysis at 72 h; Test type: Superiority; p = 0.9632, Log Rank; Difference in event probability = -0.0179, 95% CI 2-sided [-0.2143 to 0.1785]

6. Secondary Outcome: Number of Patients Dead Within 30 Days Post-transplant
Description: Mortality, defined as any death occurring in the first 30 days post-transplant, regardless of hospital discharge.
Time Frame: Up to 30 days post-transplant
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
Participants | 0 | 1

7. Secondary Outcome: Pulmonary Function Tests (FEV1=Forced Expiratory Volume in One Second and FVC=Forced Vital Capacity) at Month 1, 6 and 12 Post-transplant Evaluated According to Estenne et al.(2002).
Description: Forced expiratory volume in 1 second (FEV1) measured the amount/ volume, exhaled by a patient in the first second of the expiration after a full inspiration. Average values in healthy patients aged 20-60 range from 4.5 to 3.5 liters in males and from 3.25 to 2.5 liters in females. Forced vital capacity (FVC) was the volume of air that a patient could exhale with a maximal forced expiration effort after a deep inhaling, simply put, how much air a patient could breathe out by blowing as fast as possible. Average values in healthy patients aged 20-60 range from 5.5 to 4.75 liters in males and from 3.75 to 3.25 liters in females. The lower the values fo both parameters, the worse the outcome.
Time Frame: At months 1, 6 and 12 post-transplant
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
Litres
  FEV1 - Month 1 post transplant: number analyzed (Participants) | 38 | 42
  FEV1 - Month 1 post transplant | 2.20 (0.74) | 2.05 (0.84)
  FEV1 - Month 6 post transplant: number analyzed (Participants) | 46 | 48
  FEV1 - Month 6 post transplant | 2.62 (0.95) | 2.34 (0.85)
  FEV1 - Month 12 post transplant: number analyzed (Participants) | 45 | 46
  FEV1 - Month 12 post transplant | 2.52 (1.07) | 2.22 (0.95)
  FVC - Month 1 post transplant: number analyzed (Participants) | 38 | 42
  FVC - Month 1 post transplant | 2.49 (0.70) | 2.56 (1.01)
  FVC - Month 6 post transplant: number analyzed (Participants) | 46 | 48
  FVC - Month 6 post transplant | 3.19 (0.93) | 3.11 (0.99)
  FVC - Month 12 post transplant: number analyzed (Participants) | 45 | 46
  FVC - Month 12 post transplant | 3.19 (1.05) | 3.07 (1.10)

8. Secondary Outcome: Number of Patients With Different Bronchiolitis Obliterans Syndrome (BOS) Scores (0-3) Assessed at Months 6 and 12 Post-transplant
Description: BOS is defined as an irreversible decline in forced expiratory volume in 1 second (FEV1) of at least 20% from baseline. Spirometric measurements must be made with equipment that conforms to the American Thoracic Society standards for spirometric testing. Here the classification where stage 3 is the worst:
  BOS 0 FEV1 >90% of baseline and FEF25-75 >75% of baseline. BOS 0-p FEV1 >81% to 90% of baseline and/or FEF25-75 > 75% of baseline. BOS 1 FEV1 >66% to 80% of baseline. BOS 2 FEV1 >51% to 65% of baseline BOS 3 FEV1 >50% or less of baseline. CRF data are reported.
Time Frame: At Months 6 and 12 post-transplant
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant. Note that Out of 101 patients who entered the trial, 46 and 52 patients completed Month 1 follow-up in the repertaxin and placebo groups, respectively, and were included in the ITT population for Month 12 analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 52
Participants
  Month 6 Post Transplant - BOS Missing | 0 | 4
  Month 6 Post Transplant - BOS 0 | 45 | 44
  Month 6 Post Transplant - BOS 1 | 1 | 3
  Month 6 Post Transplant - BOS 2 | 0 | 1
  Month 6 Post Transplant - BOS 3 | 0 | 0
  Month 12 Post Transplant - Missing | 4 | 7
  Month 12 Post Transplant - BOS 0 | 35 | 36
  Month 12 Post Transplant - BOS 1 | 1 | 5
  Month 12 Post Transplant - BOS 2 | 3 | 2
  Month 12 Post Transplant - BOS 3 | 3 | 2

9. Secondary Outcome: Number of Patients With at Least One Acute Rejection Episode at Months 1, 6 and 12 Post-transplant
Description: Acute rejection was diagnosed according to Yousem et al. (1996). Histopathologic assessment of transbronchial biopsies first required confirmation of the diagnosis of mild (ACR; A2) using criteria defined in the Working Formulation for Lung Allograft Rejection. Morphological variables assessed included: one or more perivascular infiltrates in the total transbronchial biopsy fragments obtained at one bronchoscopy session, the presence of large or small airway inflammation, endothelialitis, eosinophils, plasma cells, intra-airway and intra-airspace granulation tissue, and alveolar hemosiderosis.
  The Working Formulation for grading of acute rejection of lung allografts contains five acute rejection grades:
  A0, none; A1, minimal; A2, mild; A3, moderate; and A4, severe; and is based on the intensity of perivascular mononuclear infiltrates and their extension into alveolar septa.
Time Frame: At months 1, 6 and 12 post-transplant
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
Participants
  Month 1 Post transplant | 17 | 19
  Month 6 Post Transplant | 35 | 33
  Month 12 Post Transplant | 17 | 13

10. Secondary Outcome: Patient Survival up to 12 Months Post-transplant
Description: Patient survival is derived from the date of ICU admission untile the date of death or study completion/withdrawal.
  Here this parameter is expressed as the "cumulative number of events (death)" at different timepoints till month 12, per arm.
Time Frame: at Months 3, 6, 9 and 12 post-transplant
Population: The ITT population consisted of all randomized patients who received any study medication and a lung transplant.
Measure: Number; unit: number of events
Arm/Group | Repertaxin (ITT) | Placebo (ITT)
Number analyzed (Participants) | 46 | 55
number of events
  3 Months: number analyzed (Participants) | 46 | 50
  3 Months | 0 | 3
  6 Months: number analyzed (Participants) | 46 | 48
  6 Months | 0 | 5
  9 Months: number analyzed (Participants) | 46 | 47
  9 Months | 0 | 6
  12 Months: number analyzed (Participants) | 46 | 43
  12 Months | 0 | 7
Statistical Analysis 1: Comparison: Repertaxin (ITT) vs Placebo (ITT); Herein analysis up to month 3 was reported; Test type: Superiority; p = 0.0111, Log Rank; Difference in event probability = -0.0566, 95% CI 2-sided [-0.1188 to 0.0056]
Statistical Analysis 2: Comparison: Repertaxin (ITT) vs Placebo (ITT); Herein analysis up to month 6 was reported; Test type: Superiority; p = 0.0111, Log Rank; Difference in event probability = -0.0943, 95% CI 2-sided [-0.1730 to -0.0156]
Statistical Analysis 3: Comparison: Repertaxin (ITT) vs Placebo (ITT); Herein analysis up to month 9 was reported; Test type: Superiority; p = 0.0111, Log Rank; Difference in event probability = -0.1132, 95% CI 2-sided [-0.1985 to -0.0279]
Statistical Analysis 4: Comparison: Repertaxin (ITT) vs Placebo (ITT); Herein analysis up to month 12 was reported; Test type: Superiority; p = 0.0111, Log Rank; Slope = -0.1334, 95% CI 2-sided [-0.2254 to -0.0413]

11. Secondary Outcome: Number of Patients With at Least One Adverse Events Within the First Month
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: to month 1
Population: The safety population that consisted of all patients who received any study medication and was based on the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Repertaxin (SAF) | Placebo (SAF)
Number analyzed (Participants) | 46 | 55
Participants
  Number (%) of patients reporting at least one TEAE | 46 | 55
  Number (%) of patients reporting at least one TEAE leading to discontinuation of study drug | 1 | 0
  Number (%) of patients reporting at least one serious TEAE | 14 | 14
  Number (%) of patients reporting at least one TEAE leading to death | 0 | 0
  Number (%) of patients reporting TEAEs with no relationship to study drug | 19 | 26
  Number (%) of patients reporting TEAEs with unlikely relationship to study drug | 18 | 22
  Number (%) of patients reporting TEAEs with possible study drug | 9 | 7
  Number (%) of patients reporting TEAEs with probable relationship to study drug | 0 | 0
  Number (%) of patients reporting TEAEs with highly probable relationship to study drug | 0 | 0
  Number (%) of patients reporting Serious TEAEs with no relationship to study drug | 5 | 6
  Number (%) of patients reporting Serious TEAEs with unlikely relationship to study drug | 5 | 6
  Number (%) of patients reporting Serious TEAEs with possible relationship to study drug | 4 | 2
  Number (%) of patients reporting Serious TEAEs with probable relationship to study drug | 0 | 0
  Number (%) of patients reporting Serious TEAEs with highly probable relationship to study drug | 0 | 0

12. Secondary Outcome: Number of Patients With at Least One Adverse Events From Month 1 to Month 12
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: from month 1 to month 12
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Repertaxin (SAF) | Placebo (SAF)
Number analyzed (Participants) | 46 | 52
participants
  Number of patients with TEAEs | 46 | 40
  Number (%) of patients reporting at least one TEAE | 21 | 20
  Number (%) of patients reporting at least one TEAE leading to discontinuation of study drug | 0 | 0
  Number (%) of patients reporting at least one serious TEAE | 0 | 0
  Number (%) of patients reporting at least one TEAE leading to death | 0 | 0
  Number (%) of patients reporting TEAEs with no relationship to study drug | 11 | 9
  Number (%) of patients reporting TEAEs with unlikely relationship to study drug | 9 | 8
  Number (%) of patients reporting TEAEs with possible relationship to study drug | 1 | 3
  Number (%) of patients reporting TEAEs with probable relationship to study drug | 0 | 0
  Number (%) of patients reporting TEAEs with highly probable relationship to study drug | 0 | 0

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse events data were collected was from the start of infusion to Month 12 visit. Note that in Placebo population the number of subject was 52 instead of 55 in the period from Month 1 to Month 12.
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Groups:
- Placebo (SAF): Both repertaxin and placebo were aqueous solutions packaged into identical clear glass Type I ampoule single dose units. The dosing solution for infusion was prepared aseptically at the designated Pharmacy within each center and dispensed as 12.65 mg/mL solution in appropriate size infusion bags. ampoule contained 10 mL of either repertaxin or placebo. An initial 'loading dose' of 9 mg/ml sodium chloride (NaCl) solution was administered over 30 minutes, followed by a maintenance dose lasting 47.5 hours.
  Placebo: An initial 'loading dose' of placebo was administered over 30 minutes by intravenous infusion followed by a maintenance dose lasting 47.5 hours.The infusion was to start approximately 2 hours prior to the anticipated time of reperfusion and was to continue during the ICU/hospital stay. The placebo was administered as a continuous intravenous infusion into a (high flow) central vein, by an infusion pump adequate to provide reliable infusion rates , as per treatment schedule. Total infusion volume was not to exceed 500 mL/24 hours.
  Out of 101 patients who entered the trial, 46 and 52 patients completed Month 1 follow-up in the repertaxin and placebo groups, respectively, and were included in the ITT population for Month 12 analysis. The same patients comprised the safety population. Six patients were withdrawn from the placebo group after Month 1 due to death. The same population comprised the safety population.
Arm/Group | Repertaxin (SAF) | Placebo (SAF)
All-Cause Mortality (participants affected / at risk) | 1/46 | 6/55
Serious Adverse Events (participants affected / at risk) | 14/46 | 14/55
Other Adverse Events (participants affected / at risk) | 46/46 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Repertaxin (SAF) (N=46) | Placebo (SAF) (N=55)
Coagulopathy (Blood and lymphatic system disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Lung transplant rejection (Immune system disorders) | 1 | 2
Cytokine release Syndrome (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural haemorrage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrage (Vascular disorders) | 2 | 3
Hypotension (Vascular disorders) | 0 | 3
Reperfusion injury (Vascular disorders) | 0 | 2
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Repertaxin (SAF) (N=46) | Placebo (SAF) (N=55)
Anaemia (Blood and lymphatic system disorders) | 13 | 5
Coagulopathy (Blood and lymphatic system disorders) | 4 | 3
Thromobocytopenia (Blood and lymphatic system disorders) | 3 | 4
Leukocytosis (Blood and lymphatic system disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 9 | 8
Tachycardia (Cardiac disorders) | 9 | 7
Arrhythmia (Cardiac disorders) | 3 | 3
Supraventricular tachycardia (Cardiac disorders) | 4 | 1
Atrial flutter (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 2 | 2
Pericarditis (Cardiac disorders) | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Low cardiac output syndrome (Cardiac disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0
Pericardial rub (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 28 | 21
Nausea (Gastrointestinal disorders) | 20 | 19
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 1
Abdominal distention (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 9
Pain (General disorders) | 6 | 12
Chest pain (General disorders) | 4 | 7
Oedema (General disorders) | 3 | 7
Oedema peripheral (General disorders) | 5 | 2
Fatigue (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 2
Catheter site pain (General disorders) | 1 | 1
Axillary pain (General disorders) | 1 | 0
Bloody discharge (General disorders) | 0 | 1
Catheter related complication (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Local swelling (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Lung transplant rejection (Immune system disorders) | 2 | 2
Cytokine release syndrome (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 3
Pseudomonas infection (Infections and infestations) | 2 | 2
Staphylococcal infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 0 | 2
Aspergillosis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 2
Enterobacter infection (Infections and infestations) | 1 | 0
Enterobacter pneumonia (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 1
Klebisiella infection (Infections and infestations) | 0 | 1
Laryngotracheo bronchitis (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Mycoplasma infection (Infections and infestations) | 2 | 0
Nocardiosis (Infections and infestations) | 0 | 1
Pneumonia Klebisiella (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Upper repiratory fungal infection (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 35 | 33
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Thrombosis in device (Injury, poisoning and procedural complications) | 2 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 1
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Device failure (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 2
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Liver function test abnormal (Investigations) | 5 | 3
Haematocrit decreased (Investigations) | 2 | 4
White blood cell count increased (Investigations) | 1 | 5
Blood creatinine increased (Investigations) | 4 | 1
Blood phosphorus decreased (Investigations) | 3 | 1
Urine output decreased (Investigations) | 1 | 3
Blood magnesium decreased (Investigations) | 2 | 1
Blood potassium decreased (Investigations) | 1 | 2
Oxygen saturation decreased (Investigations) | 1 | 2
Electrocardiogram ST segment elevation (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Cardiac output decreased (Investigations) | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 2
Electrocardiogram abnormal (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1
Respiratory rate decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Urine output increased (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 13
Hypovolaemia (Metabolism and nutrition disorders) | 7 | 13
Hypervolaemia (Metabolism and nutrition disorders) | 5 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponantraemia (Metabolism and nutrition disorders) | 3 | 1
Acidosis (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydratation (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalace (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 3
Convulsion (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 2 | 0
Unresponsive to verbal stimuli (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 11 | 13
Anxiety (Psychiatric disorders) | 4 | 7
Hallucination (Nervous system disorders) | 3 | 4
Agitation (Psychiatric disorders) | 2 | 1
Restlessness (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 0 | 3
Mental status changes (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 4
Renal tubular disorder (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2
Anuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 14 | 14
Haemorrhage (Vascular disorders) | 6 | 10
Hypertension (Vascular disorders) | 5 | 6
Reperfusion injury (Vascular disorders) | 1 | 2
Haemodynamic instability (Vascular disorders) | 0 | 2
Flushing (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2006-03-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT00224406/Prot_000.pdf
  • Statistical Analysis Plan (2006-09-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT00224406/SAP_001.pdf